CLINICAL TRIAL: NCT05267977
Title: Antibiotic Use & Open Fracture of the Lower Extremity
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated by PI due to limited resources, no data collected
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 041.TRA.2016.D
Record Dates: First submitted 2019-08-12; First posted 2022-03-07 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-08

CONDITIONS: Lower Extremity Fracture
Keywords: Gustilo
MeSH Terms: interventions — First Generation Cephalosporins; Aminoglycosides

STUDY DESIGN:
Intervention Model Description: Phase: Part 1: Retrospective multi-center study. Part 2: Prospective multi-center study. Number of Sites: Methodist Health System and the associated center. Description of Intervention: Phase 1: No intervention. Phase 2: Patients will be randomized to receive either cephalosporin or the combination of cephalosporin and aminoglycoside.
  Study Duration: Phase 1: 3 years. Phase 2: 5 years. Subject Participation Duration: Phase 2: Patients will be enrolled in the study until discharge from the hospital. Study participation is strictly voluntary and patient can withdraw at any time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- cephalosporin (Active Comparator): cephalosporin
  Interventions: Drug: Cephalosporin 1St Generation
- cephalosporin and aminoglycoside (Active Comparator): the combination of cephalosporin and aminoglycoside.
  Interventions: Drug: Cephalosporin 1St Generation; Drug: Aminoglycosides

INTERVENTIONS:
Drug: Cephalosporin 1St Generation
Drug: Aminoglycosides
  Arms: cephalosporin and aminoglycoside

SUMMARY:
It is important to recognize the potential for renal injury and be cognizant of this during the management of complex trauma patients. The primary aim of this study is to investigate the necessity of aminoglycoside usage for patients with open lower extremity fractures. Hypothesis: adding aminoglycoside on top of cephalosporin in treating lower extremity fracture will make no significant difference in term of clinical outcomes when compared to cephalosporin alone.

DETAILED DESCRIPTION:
The trauma patient is particularly susceptible to renal injury due to factors such as renal hypoperfusion in the acute setting, the concomitant administration of necessary intravenous contrast agents for diagnostic, and sometimes additionally therapeutic imaging (3). This is additionally complicated by the presentation of trauma patients with pre-existing renal disease.

This study will assess whether prophylactic antibiotics <72hrs have similar outcomes as ≥ 72 hrs of antibiotics, whether type of antibiotics impacts outcomes in patients in either group, help determine the incidence of infection in Gustilo Type III lower extremity fracture when treated either with a single agent (cephalosporin) or dual agent (cephalosporin + aminoglycoside) and the complication profile of patients with Gustilo Type III lower extremity fracture when treated either with a single agent (cephalosporin 1st generation) or dual agent (cephalosporin 1st generation + aminoglycoside).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years of age
* All patients with open grade II or grade III lower extremity open fractures according to the Gustilo Classification of open fracture.

Exclusion Criteria:

* Any significant injuries in addition to the lower extremity fracture as determined by the PI that may confound the data.
* Inability to give informed consent or comply with data acquisition (Part 3).
* Pregnant or breast feeding patients due to the potential risks to the mother and/or fetus.
* Prisoners
* Previous bone malignancy
* Bowel or enteric injury at index admission
* TBI of AIS ≥ 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Aminoglycoside Usage | Within 24 hours of admission
  The necessity of aminoglycoside usage for patients with open lower extremity fractures.

SECONDARY OUTCOMES:
Demographics | Within 24 hours of admission
  age, sex, ethnicity
comorbidities | Within 24 hours of admission
  in regards to necessity of aminoglycoside usage for patients with open lower extremity fractures
Total hospital length of stay - HLOS | Within 24 hours of admission
  in regards to necessity of aminoglycoside usage for patients with open lower extremity fractures
deep space infection (DSI) | Within 24 hours of admission
  in regards to necessity of aminoglycoside usage for patients with open lower extremity fractures
grade of fracture | Within 24 hours of admission
  in regards to necessity of aminoglycoside usage for patients with open lower extremity fractures
surgical site infection (SSI) | Within 24 hours of admission
  in regards to necessity of aminoglycoside usage for patients with open lower extremity fractures

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Truitt, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Health System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No